CLINICAL TRIAL: NCT05193513
Title: Comparison of Tow Maxillary Hybrid Expanders -Perpendicular Screw Supported Versus Lateral Angulated One; a Prospective Randomized Clinical Study
Brief Title: Tow Maxillary Hybrid Expanders Screw Supported Versus Lateral Angulated One; a Prospective Randomized Clinical Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Abdallah EL sayed Mohamed Hassan, Comparison of tow maxillary hybrid expanders -perpendicular screw Supported versus lateral angulated one; a prospective randomized clinical study, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 628/3133
Record Dates: First submitted 2022-01-03; First posted 2022-01-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Cross Bite
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group (1) (Experimental): tow perpendicular miniscrews supported hybrid expanders
  Interventions: Device: hybrid expanders
- group (2) (Experimental): tow angulated miniscrews supported hybrid expanders
  Interventions: Device: hybrid expanders

INTERVENTIONS:
Device: hybrid expanders — tow maxillary hybrid expanders supported anteriorly with tow miniscrews

SUMMARY:
in this study i will use to different designs of t maxillary hybrid expanders that consists of HYREX supported with tow miniscrews to treat the collapsed maxilla in Yonge adolescents

DETAILED DESCRIPTION:
the maxilla is expanded by tow diffrent designs of maxillary hybrid expanders

ELIGIBILITY:
Inclusion Criteria:

1. Medically free male or female patients
2. Patients that necessitated maxillary expansion due to constricted maxillary arch shown by a unilateral or bilateral posterior crossbite.
3. The patient should have no missing teeth except third molars.
4. Age ranged from 12 to 18 years old.
5. The patient should have a good gingival condition.
6. The patient should have a good periodontal condition.

Exclusion Criteria:

1-hisory of previous orthodontic treatment. 2- Lack of cooperation. 3- Mental problems. 4- Skeletal open bite. 5- TMJ problem.

-

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2021-07-10 (Actual); Primary Completion 2023-06-10 (Estimated); Study Completion 2023-10-14 (Estimated)

PRIMARY OUTCOMES:
change in maxillary width | 12 weeks following end of treatment
  millimeter

CONTACTS AND LOCATIONS:
Locations (1):
- Al azhar university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided